CLINICAL TRIAL: NCT01943851
Title: A Phase I/II Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK525762 in Subjects With Relapsed, Refractory Hematologic Malignancies
Brief Title: A Dose Escalation Study to Investigate the Safety, Pharmacokinetics (PK), Pharmacodynamics (PD) and Clinical Activity of GSK525762 in Subjects With Relapsed, Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116183; 2013-000445-39 (EudraCT Number)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms
Keywords: leukemia; Acute myeloid leukemia; BET inhibitor; lymphoma; Myelodysplastic syndromes; Oncology; multiple myeloma; GSK525762
MeSH Terms: conditions — Neoplasms; Leukemia; Leukemia, Myeloid, Acute; Lymphoma; Myelodysplastic Syndromes; Multiple Myeloma | interventions — molibresib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: GSK525762 QD Cohort (Experimental): Subject will be administered a 5 milligram (mg) starting dose of GSK525762, oral tablets, QD. Dose escalations will be performed in Part 1 and dose adjustments are allowed to address tolerability and safety issues. Thereafter, subjects will be enrolled in a standard 3+3 design. Separate dose escalation cohorts will be opened for subjects with AML, NHL, and MM for QD dosing. Dose escalation will continue until an MTD is determined or until a dose of 200 mg per day is reached.
  Interventions: Drug: GSK525762
- Part 1: GSK525762 BID Cohort (Experimental): Subject will be administered a starting dose of GSK525762, oral tablets, 20 mg BID (12 hours apart, total daily dose of 40 mg). Dose escalations will be performed in Part 1 and dose adjustments are allowed to address tolerability and safety issues. Thereafter, subjects will be enrolled in a standard 3+3 design. Separate dose escalation cohorts will be opened for subjects with AML, NHL, and MM, for BID dosing. Dose escalation will continue until an MTD is determined or until a dose of 200 mg per day is reached.
  Interventions: Drug: GSK525762
- Part 2: GSK525762 dose expansion cohort (Experimental): After the MTD has been determined in Part1, Part 2 dose expansion cohorts will be opened for AML, NHL and MM.
  Interventions: Drug: GSK525762

INTERVENTIONS:
Drug: GSK525762 — GSK525762 1 mg, 10 mg and 30 mg will be supplied as white to off-white, amorphous free base and white to slightly colored crystalline besylate tablets, round, biconvex tablets with no markings. GSK525762 will be administered with 240 milliliter (mL) water.

SUMMARY:
This is an open-label repeat dose, multicenter, 2-part study to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) for GSK525762 given once-daily (QD) orally. Part 1 of the study is a dose escalation phase to select the recommended Part 2 dose (RP2D) based on the safety, PK, and PD profiles observed after oral administration of GSK525762. Eligible subjects with select relapsed refractory hematological malignancies (acute myeloid leukemia [AML], non-Hodgkin's Lymphoma [NHL]and multiple myeloma [MM]), will be enrolled in the QD and/or BID dosing cohorts until a MTD is established. Subjects may continue treatment in the study until disease progression, unacceptable toxicity, or withdrawal of consent. . Upon determination of the MTD, twice daily (BID) dosing cohorts may be opened to collect additional safety data and evaluate the preliminary efficacy of GSK525762 administered BID. Part 2 will explore clinical activity at the MTD or RP2D; separate expansion cohorts will be planned for acute myeloid leukemia (AML), non-Hodgkin's Lymphoma (NHL, including an exploratory sub-cohort of subjects with myc and B-Cell Leukemia (BCL)2 and/or BCL6 rearrangements/overexpression [double- and triple-hit lymphoma]), and multiple myeloma (MM). This is the first study of this agent to be conducted in subjects with these relapsed and/or refractory hematological malignancies for which no standard therapies are anticipated to result in a durable remission.

ELIGIBILITY:
Inclusion criteria

* Written informed consent provided.
* Males and females 18 years old or older.
* In Part 1 and, Part 2, subjects must have AML, MM, or NHL. Subjects with AML, are eligible if they • have relapsed and/or refractory disease, OR are>=65 years of age and not candidates for or have refused standard chemotherapy. Subjects with multiple myeloma are eligible if they have progressed despite therapy with an alkylating agent, proteasome inhibitor, and immunomodulatory agent, either as individual regimens or in combination. Subjects with NHL are eligible if they have received at least two prior lines of systemic therapy, including at least one line of immunochemotherapy with an anti-CD20 antibody (if their tumor expresses CD20).

In Part 2, the NHL cohort will separately enrol subjects with double- and triple hit lymphoma, so that a minimum of 10 subjects with this subset of disease will be enrolled. To be eligible for this sub-cohort, tumor sample from the subject must demonstrate rearrangement and/or overexpression of MYC and either BCL2 and/or BCL6 genes. Evaluation of double- or triple-hit status may be performed via appropriate local testing, and the determination of double- or triple-hit diagnosis will be at the discretion of the investigator and GSK Medical Monitor.

* Subjects with a prior history of stem cell transplant (autologous and/or allogeneic) are allowed if

  * At least 3 months has elapsed from the time of transplant and
  * the subject has recovered from transplant-associated toxicities prior to the first dose of GSK525762, and For subjects with a prior history of allogeneic transplant,
  * the subject has been off systemic immunosuppressive medications (including but not limited to: cyclosporine, tacrolimus, mycophenolate mofetil, or corticosteroids) for at least 1 month prior to the first dose of GSK525762. Topical steroids are permitted
  * there are no signs or symptoms of graft versus host disease, other than Grade 1 skin involvement.
* Eastern Cooperative Oncology Group (ECOG) performance status of <=1.
* Subject must be stable enough to be expected to complete dosing through the DLT observation period as assessed by the investigator.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-International units per milliliter and estradiol < 40 picograms per milliliter (< 140 picomole per liter) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods defined in protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least two to four weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until at least 7 months after the last dose of study medication; Negative serum pregnancy test <= 7 days prior to first study drug dose; Female subjects who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for 5 half-lives of GSK525762 or at least 28 days (whichever is longer) following the last dose of study treatment.
* Male subjects must agree to use one of the methods of contraception specified. This method must be used from the time of the first dose of study medication until 16 weeks after the last dose of study medication. In addition, male subjects whose partners are or become pregnant must continue to use condoms for 7 days after stopping study medications.
* Adequate organ system function.
* Ability to comply with dietary and tobacco/alcohol abstinence requirements.

Exclusion Criteria

* Haematological malignancy associated with human immunodeficiency virus (HIV) infection or solid organ transplant or history of known Hepatitis B Antigen or positive Hepatitis C antibody (confirmed by Recombinant ImmunoBlot Assay [RIBA], if available or alternately confirmed by Hepatitis C Virus [HCV] Ribonucleic acid [RNA]).
* History or concurrent malignancy of solid tumours, except for below. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled even if less than 5 years have elapsed since treatment. Consult the GSK Medical Monitor if unsure whether second malignancies meet requirements specified above.
* Currently receiving cancer therapy (chemotherapy, radiation therapy, immuno- therapy, biologic therapy, hormonal therapy, surgery, and/or tumour embolization).The following are allowed: Hydroxyurea for proliferative disease, Corticosteroids, Use of hematopoetic growth factors is permitted at the discretion of the investigator according to published guidelines (e.g., National Comprehensive Cancer Network (NCCN), American Society of Clinical Oncology (ASCO), American Society of Hematology (ASH), etc.). The following are NOT allowed: Investigational anti cancer drug within 2 weeks prior to the first dose of GSK525762; Major surgery, radiotherapy, or immunotherapy within 4 weeks of GSK525762 Chemotherapy regimens with delayed toxicity within the last 4 weeks. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.

Nitrosourea or mitomycin C within the last 6 weeks

* Evidence of severe of uncontrolled infection.
* Use of anticoagulants (e.g., warfarin, heparin) at therapeutic levels within 7 days prior to the first dose of GSK525762. Low dose (prophylactic) low molecular weight heparin (LMWH) is permitted. In addition, INR must be monitored in accordance with local institutional practices, as appropriate.
* Current use of a prohibited medication or requires any of these medications during treatment with the investigational drugs. This includes excluding current medications known or suspected to be associated QT prolongation. In addition, any subject who is expected to require a QT prolonging medication while on trial should not be enrolled.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator.
* Symptomatic or untreated Central nervous system (CNS) disease, Subjects with a history of CNS disease (leukemia, lymphoma or myeloma) are permitted to enrol if they have previously received appropriate therapy and CNS remission has been documented. Subject with primary CNS lymphoma (defined as isolated CNS lymphoma without systemic involvement) are excluded from study.
* Cardiac abnormalities as evidenced by any of the following: History or current clinically significant uncontrolled arrhythmias or hypertension; Clinically significant conduction abnormalities or arrhythmias, subjects with Bundle Branch Block; Presence of cardiac pacemaker; History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months.
* Any of the following ECG findings or assessments including: Baseline QTcF interval >=450 milliseconds; Clinically significant ECG assessments should be reviewed by the site cardiologist prior to study entry.
* GSK525762 is a benzodiazepine class molecule. Any serious known immediate or delayed hypersensitivity reaction(s) to GSK525762 or idiosyncrasy to drugs chemically related to the investigational drug.
* Evidence of hemoptysis within the last 7 days.
* History of major gastrointestinal bleeding within the last 3 months or any evidence of active gastrointestinal bleeding excludes the subject.
* Presence of gastrointestinal disease that would significantly affect compound absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (5):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, East Melbourne, Victoria, Australia
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Salamanca
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Bell C; Fennell K; Chan YC; Rambow F; Yeung M; Vassiliadis D; Lara L; Yeh P; Martelotto L; Rogiers A; Kremer B; Barbash O; Mohammad H; Johanson T; Burr M; Dhar A; Karpinich N; Tian L; Tyler D; MacPherson L; Shi J; Pinnawala N; Fong CY; Papenfuss A; Grimmond S; Dawson SJ; Allan R; Kruger R; Vakoc C; Goode D; Naik S; Gilan O; Lam E; Marine JC; Prinjha R; and Dawson M.Enhancer remodeling overcomes therapeutic resistance driven by epigenetic evolution in cancer.Nature.2019;
- [Derived] Dawson MA, Borthakur G, Huntly BJP, Karadimitris A, Alegre A, Chaidos A, Vogl DT, Pollyea DA, Davies FE, Morgan GJ, Glass JL, Kamdar M, Mateos MV, Tovar N, Yeh P, Delgado RG, Basheer F, Marando L, Gallipoli P, Wyce A, Krishnatry AS, Barbash O, Bakirtzi E, Ferron-Brady G, Karpinich NO, McCabe MT, Foley SW, Horner T, Dhar A, Kremer BE, Dickinson M. A Phase I/II Open-Label Study of Molibresib for the Treatment of Relapsed/Refractory Hematologic Malignancies. Clin Cancer Res. 2023 Feb 16;29(4):711-722. doi: 10.1158/1078-0432.CCR-22-1284. PMID 36350312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label repeat dose, multicenter study to investigate the safety, pharmacokinetics (PK), pharmacodynamics and clinical activity of GSK525762 in participants with relapsed, refractory hematologic malignancies. The study was conducted in 2 parts: Part 1 (dose escalation) and Part 2 (dose expansion)
Pre-assignment Details: A total of 111 participants were enrolled (87 participants in Part 1 and 24 participants in Part 2) across the study centers in Australia, Spain, Great Britain, South Korea and United State of America (USA).
Groups:
- Part 1: GSK525762 5 mg QD: Participants were administered once daily oral dose of 5 milligrams (mg) GSK525762.
- Part 1: GSK525762 10 mg QD: Participants were administered once daily oral dose of 10 mg GSK525762.
- Part 1: GSK525762 20 mg QD: Participants were administered once daily oral dose of 20 mg GSK525762.
- Part 1: GSK525762 30 mg QD MM: Participants with multiple myeloma (MM) were administered once daily oral dose of 30 mg GSK525762.
- Part 1: GSK525762 40 mg QD: Participants were administered once daily oral dose of 40 mg GSK525762.
- Part 1: GSK525762 40 mg QD MM: Participants with MM were administered once daily oral dose of 40 mg GSK525762.
- Part 1: GSK525762 60 mg QD AML: Participants with Acute Myeloid Leukemia (AML) were administered once daily oral dose of 60 mg GSK525762.
- Part 1: GSK525762 60 mg QD NHL: Participants with Non-Hodgkin's Lymphoma (NHL) were administered once daily oral dose of 60 mg GSK525762.
- Part 1: GSK525762 60 mg QD MM: Participants with MM were administered once daily oral dose of 60 mg GSK525762.
- Part 1: GSK525762 75 mg QD AML: Participants with AML were administered once daily oral dose of 75 mg GSK525762.
- Part 1: GSK525762 80 mg QD: Participants were administered once daily oral dose of 80 mg GSK525762.
- Part 1: GSK525762 80 mg QD AML: Participants with AML were administered once daily oral dose of 80 mg GSK525762.
- Part 1: GSK525762 80 mg QD NHL: Participants with NHL were administered once daily oral dose of 80 mg GSK525762.
- Part 1: GSK525762 100 mg QD AML: Participants with AML were administered once daily oral dose of 100 mg GSK525762.
- Part 1: GSK525762 120 mg QD AML: Participants with AML were administered once daily oral dose of 120 mg GSK525762.
- Part 2: GSK525762 60 mg QD CTCL: Participants Cutaneous T cell lymphoma (CTCL) were administered once daily oral dose of 60 mg GSK525762.
- Part 2: GSK525762 75 mg QD MDS: Participants with Myelodysplastic Syndrome (MDS) were administered once daily oral dose of 75 mg GSK525762.
- Part 2: GSK525762 80 mg QD CTCL: Participants CTCL were administered once daily oral dose of 80 mg GSK525762
Period: Part 1 (Up to 86.9 Weeks)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Started | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 4 | 0 | 4 | 7 | 16 | 2 | 8 | 1 | 7 | 7 | 15 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 36.4 Weeks)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 16 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 13 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Population: NA indicates, Data not presented due to participant confidentiality and privacy concerns
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL | Total
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6 | 7 | 16 | 1 | 111
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 1 | 0 | 0 | 4 | 0 | 3 | 3 | 11 | 3 | 3 | 0 | 3 | 4 | 7 | 4 | 4 | 1 | 0 | 51
  65-74 years | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 5 | 0 | 3 | 0 | 2 | 3 | 3 | 1 | 2 | 9 | 1 | 36
  >74 years | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 6 | 1 | 1 | 6 | 0 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 2 | NA — Data not presented due to patient confidentiality and privacy concerns | 2 | 1 | 5 | 1 | 7 | NA — Data not presented due to patient confidentiality and privacy concerns | 4 | 2 | 6 | 1 | 5 | 6 | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 3 | NA — Data not presented due to patient confidentiality and privacy concerns | 2 | 7 | 13 | 2 | 1 | NA — Data not presented due to patient confidentiality and privacy concerns | 3 | 5 | 10 | 5 | 2 | 10 | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese Heritage(H)/eastAsian (H)/Southeast Asian (H) | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 2 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 5 | 1 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 1 | 1 | 0 | 1 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African american | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 1 | 1 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 2 | 0 | 0 | 0 | 0 | 1 | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native hawaiian or other pacific islander | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 0 | 0 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 1 | 0 | 0 | 0 | 0 | NA — NA indicates, Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 3 | NA — Data not presented due to patient confidentiality and privacy concerns | 4 | 6 | 12 | 1 | 8 | NA — Data not presented due to patient confidentiality and privacy concerns | 5 | 5 | 14 | 6 | 5 | 15 | NA — NA indicates, Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian and native hawaiian or other pacific islander | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 0 | 0 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 0 | 0 | 0 | 0 | NA — NA indicates, Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.
  Missing | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 2 | 0 | 0 | 0 | NA — Data not presented due to patient confidentiality and privacy concerns | 0 | 0 | 1 | 0 | 1 | 0 | NA — NA indicates, Data not presented due to patient confidentiality and privacy concerns | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) and AE Leading to Discontinuation (AELD)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and SAE is defined as any untoward medical occurrence that, at any dose which results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or, is a congenital anomaly/birth defect. AELD is adverse events leading to permanent discontinuation of study treatment.
Time Frame: Up to 86.9 weeks
Population: All Treated Population consists of all participants that received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  Non-serious AEs | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  SAEs | 1 | 0 | 0 | 4 | 0 | 3 | 6 | 12 | 2 | 8 | 1 | 6 | 7 | 14 | 6
  AELD | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 0 | 2 | 0 | 3 | 1 | 8 | 2

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: An event was considered DLT if it occurred within first 3weeks of treatment & met one of following criteria:unless it was clearly established that event is unrelated to treatment:Grade4 neutropenia persisting for >=7 days/febrile neutropenia not responding to treatment within 24hours, Grade4 thrombocytopenia lasting more than 7day & not responding to transfusions/Grade3 thrombocytopenia associated with bleeding (>10milliliter [mL]), Drug-related Grade 3/4 non-hematologic toxicity as described in National Cancer Institute-Common Terminology Criteria for Adverse Events(NCI-CTCAE)version 4.0, Drug-related Grade2 non-hematological toxicity, Grade2 Troponin T elevation(central laboratory>Upper Limit of Normal[ULN]),measured on two separate occasions within 48 hours, Treatment delay of 14 days/greater due to unresolved drug-related toxicity,ALT>=3xULN+bilirubin>=2xULN(>35% direct)/Alanine aminotransferase(ALT) between 3-5xULN with bilirubin<2xULN but with hepatitis symptom/rash/ALT>=5xULN.
Time Frame: Up to 3 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: GSK525762 40 mg QD MM: Participants with multiple myeloma were administered once daily oral dose of 40 mg GSK525762.
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Part 1: Number of Participants With Dose Reductions
Description: Number of participants with dose reductions due to any reason is presented.
Time Frame: Up to 86.9 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | 1 | 0 | 0 | 5 | 3 | 1

4. Primary Outcome: Part 1: Number of Participants With Any Dose Interruptions or Delays
Description: Number of participants with any dose interruptions/ delays is presented.
Time Frame: Up to 86.9 weeks
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants | 1 | 0 | 1 | 3 | 0 | 3 | 5 | 15 | 2 | 7 | 1 | 6 | 7 | 13 | 6

5. Primary Outcome: Part 1: Number of Participants With Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: glucose, prothrombin international normalized ratio (Pro. INR), albumin, amylase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, calcium, calcium ionized, cholesterol, creatinine, creatine kinase, lipase, potassium, magnesium, sodium, triglycerides, alkaline phosphatase (ALP). Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Higher grade indicates greater severity. An increase was defined as an increase relative to Baseline. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post Baseline with any grade increase is presented.
Time Frame: Up to 86.9 weeks
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  Glucose, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Glucose, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 1 | 0 | 1 | 3 | 1 | 3 | 6 | 16 | 2 | 8 | 1 | 6 | 6 | 15 | 3
  Pro.INR, n=0,1,1,5,1,3,4,16,3,4,0,6,5,11,4: number analyzed (Participants) | 0 | 1 | 1 | 5 | 1 | 3 | 4 | 16 | 3 | 4 | 0 | 6 | 5 | 11 | 4
  Pro.INR, n=0,1,1,5,1,3,4,16,3,4,0,6,5,11,4 |  | 0 | 1 | 3 | 0 | 1 | 3 | 10 | 1 | 3 |  | 4 | 5 | 8 | 3
  Albumin, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Albumin, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 7 | 1 | 3 | 1 | 3 | 3 | 6 | 1
  ALT, n=1,1,1,5,1,4,8,18,3,8,1,7,7,15,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 15 | 6
  ALT, n=1,1,1,5,1,4,8,18,3,8,1,7,7,15,6 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 1 | 1 | 0 | 1 | 3 | 4 | 0
  Amylase, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,5: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 5
  Amylase, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,5 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 5 | 2 | 0 | 0 | 3 | 4 | 3 | 0
  AST, n=1,1,1,5,1,4,8,18,3,8,1,7,7,16,6 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 3 | 3 | 4 | 1
  Bilirubin, n=1,1,1,5,1,4,8,18,3,8,1,7,7,16,6 | 1 | 0 | 1 | 0 | 1 | 1 | 6 | 8 | 1 | 7 | 1 | 6 | 5 | 12 | 4
  Calcium, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Calcium, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 0 | 0 | 0 | 2 | 0 | 1 | 5 | 6 | 0 | 5 | 0 | 4 | 1 | 6 | 5
  Calcium Ionized, n=1,1,1,4,1,4,7,17,3,8,1,7,7,15,6: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 7 | 17 | 3 | 8 | 1 | 7 | 7 | 15 | 6
  Calcium Ionized, n=1,1,1,4,1,4,7,17,3,8,1,7,7,15,6 | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 3 | 0 | 3 | 3 | 6 | 2
  Cholesterol,n=1,1,1,4,1,4,3,17,3,6,1,7,6,10,3: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 17 | 3 | 6 | 1 | 7 | 6 | 10 | 3
  Cholesterol,n=1,1,1,4,1,4,3,17,3,6,1,7,6,10,3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 0
  Creatine Kinase, n=1,1,1,2,1,4,8,18,3,7,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 4 | 8 | 18 | 3 | 7 | 1 | 7 | 7 | 16 | 6
  Creatine Kinase, n=1,1,1,2,1,4,8,18,3,7,1,7,7,16,6 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 2 | 4 | 0
  Creatinine, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Creatinine, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 5 | 1 | 1 | 0 | 3 | 2 | 6 | 1
  Lipase, n=1,1,1,5,1,4,6,18,3,8,1,7,6,15,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 6 | 18 | 3 | 8 | 1 | 7 | 6 | 15 | 6
  Lipase, n=1,1,1,5,1,4,6,18,3,8,1,7,6,15,6 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 0 | 2 | 0 | 2 | 3 | 0 | 1
  Potassium, n=1,1,1,5,1,4,7,18,3,8,1,7,6,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 6 | 16 | 6
  Potassium, n=1,1,1,5,1,4,7,18,3,8,1,7,6,16,6 | 1 | 0 | 1 | 1 | 0 | 3 | 3 | 4 | 2 | 5 | 1 | 5 | 4 | 7 | 3
  Magnesium,n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Magnesium,n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 4 | 2 | 1 | 1 | 4 | 5 | 8 | 2
  Sodium, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
  Sodium, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 1 | 0 | 0 | 3 | 1 | 3 | 3 | 6 | 1 | 4 | 1 | 4 | 2 | 9 | 3
  Triglycerides, n=1,1,1,4,1,4,3,17,3,6,1,7,6,10,3: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 17 | 3 | 6 | 1 | 7 | 6 | 10 | 3
  Triglycerides, n=1,1,1,4,1,4,3,17,3,6,1,7,6,10,3 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 4 | 1 | 3 | 1 | 5 | 2 | 8 | 2
  ALP, n=1,1,1,5,1,4,8,18,3,8,1,7,7,16,6 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 4 | 3 | 1 | 1

6. Primary Outcome: Part 1: Number of Participants With Grade Change From Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Higher grade indicates greater severity. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post Baseline with any grade increase is presented.
Time Frame: Up to 86.9 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  Hemoglobin, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 1 | 0 | 0 | 2 | 0 | 2 | 3 | 13 | 3 | 6 | 1 | 4 | 6 | 9 | 3
  Lymphocytes, n=1,1,0,5,1,4,7,18,3,8,1,7,7,15,6: number analyzed (Participants) | 1 | 1 | 0 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 15 | 6
  Lymphocytes, n=1,1,0,5,1,4,7,18,3,8,1,7,7,15,6 | 0 | 0 |  | 3 | 1 | 3 | 4 | 11 | 2 | 5 | 1 | 6 | 3 | 10 | 5
  Neutrophils, n=1,1,0,5,1,4,7,18,3,8,1,7,7,15,5: number analyzed (Participants) | 1 | 1 | 0 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 15 | 5
  Neutrophils, n=1,1,0,5,1,4,7,18,3,8,1,7,7,15,5 | 0 | 0 |  | 4 | 0 | 3 | 1 | 6 | 2 | 5 | 0 | 2 | 5 | 3 | 1
  Platelets, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 0 | 0 | 1 | 4 | 1 | 4 | 4 | 17 | 3 | 4 | 1 | 5 | 7 | 11 | 2
  Leukocytes, n=1,1,1,5,1,4,7,18,3,8,1,7,7,16,6 | 0 | 0 | 1 | 4 | 1 | 3 | 2 | 9 | 3 | 4 | 1 | 3 | 4 | 9 | 3

7. Primary Outcome: Part 1: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected to assess glucose, ketones, occult blood, urine protein, and monoclonal protein (monoclonal pro). The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Any increase was defined as any increase in proportional concentrations relative to Baseline. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post Baseline with any increase is presented.
Time Frame: Up to 86.9 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 5 | 15 | 3 | 7 | 1 | 6 | 5 | 11 | 2
Participants
  Glucose, n=1,1,1,4,1,4,4,15, 3,5,0,3,5,8,1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 4 | 15 | 3 | 5 | 0 | 3 | 5 | 8 | 1
  Glucose, n=1,1,1,4,1,4,4,15, 3,5,0,3,5,8,1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 |  | 0 | 2 | 2 | 1
  Ketones, n=1,1,1,4,1,4,4,13,3,5,1,6,5,11,2: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 4 | 13 | 3 | 5 | 1 | 6 | 5 | 11 | 2
  Ketones, n=1,1,1,4,1,4,4,13,3,5,1,6,5,11,2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 3 | 1
  Occult blood, n=1,1,1,4,1,4,5,14,3,7,1,6,5,11,2: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 5 | 14 | 3 | 7 | 1 | 6 | 5 | 11 | 2
  Occult blood, n=1,1,1,4,1,4,5,14,3,7,1,6,5,11,2 | 1 | 0 | 1 | 3 | 0 | 2 | 3 | 4 | 3 | 3 | 1 | 4 | 2 | 4 | 1
  Protein, n=1,1,1,4,1,4,2,12,1,5,0,3,4,7,1: number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 2 | 12 | 1 | 5 | 0 | 3 | 4 | 7 | 1
  Protein, n=1,1,1,4,1,4,2,12,1,5,0,3,4,7,1 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 5 | 0 | 3 |  | 0 | 3 | 3 | 1
  Monoclonal pro, n=0,0,0,0,0,1,0,0,2,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Monoclonal pro, n=0,0,0,0,0,1,0,0,2,0,0,0,0,0,0 |  |  |  |  |  | 0 |  |  | 0 |  |  |  |  |  |

8. Primary Outcome: Part 1: Number of Participants With Worst Case Vital Signs Results Relative to Baseline: Pulse Rate and Body Temperature
Description: Vital signs (pulse rate and temperature) were measured after resting for at least 5 minutes in a supine or semi-recumbent position. The clinical concern ranges were: For pulse rate (low <60 beats per minute [bpm] and high >100 bpm); For body temperature (<=35 degrees Celsius or >=38 degrees Celsius). Participants were counted in the worst case category that their value changed to (low, normal or high), unless there was no change in their category. Participants whose value category was unchanged, or whose value became normal, were recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date.
Time Frame: Up to 86.9 weeks
Population: All Treated Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  Pulse rate, To Low | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pulse rate, To Normal or No change | 0 | 1 | 0 | 2 | 0 | 2 | 4 | 8 | 1 | 5 | 1 | 1 | 1 | 8 | 4
  Pulse Rate, To High | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 10 | 2 | 3 | 0 | 6 | 6 | 8 | 2
  Temperature, To Low | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Temperature, To Normal or No Change | 0 | 1 | 1 | 4 | 1 | 2 | 3 | 15 | 3 | 7 | 1 | 1 | 6 | 7 | 6
  Temperature, To High, | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 3 | 0 | 1 | 0 | 6 | 0 | 8 | 0

9. Primary Outcome: Part 1: Number of Participants With Increase to Grade 3 From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured after resting for at least 5 minutes in a supine or semi-recumbent position. They were graded according to NCI-CTCAE version 4.0. For SBP: Grade 0 (<=120 millimeter of mercury [mmHg]), Grade 1 (121-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg). For DBP: Grade 0 (<=80 mmHg), Grade 1 (81-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg). Higher grade indicates greater severity. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. An increase is defined as an increase in grade relative to Baseline grade. Number of participants with increase to Grade 3 from Baseline is presented.
Time Frame: Up to 86.9 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  DBP | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  SBP | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 4 | 1 | 4 | 4

10. Primary Outcome: Part 1: Number of Participants With Worst-case Post-Baseline Abnormal Electrocardiogram (ECG) Findings (Investigator Reading)
Description: 12-lead ECGs were recorded with the participants in a supine position using an ECG machine. Number of participants with worst-case clinically significant and not clinically significant abnormal ECG findings have been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to 86.9 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Participants
  Abnormal-Clinically significant | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 1
  Abnormal-Not Clinically significant | 1 | 1 | 0 | 4 | 1 | 3 | 6 | 17 | 3 | 5 | 1 | 7 | 5 | 12 | 5

11. Primary Outcome: Part 2: Objective Response Rate (ORR) (MDS Cohort)
Description: ORR for MDS cohort is defined as the percentage of participants achieving Complete Response (CR), Marrow CR, CRp (as per CR but platelet count <100 x 10^9 cells/Liter[L]), CRi (as per CR but platelet count <100 x 10^9cells/L or neutrophil count <1 x 10^9 cells/L), or Partial Response (PR) per response criteria. Complete response is defined as bone marrow <=5% myeloblasts with normal maturation of all cell lines, with hemoglobin concentration of >=11 grams per deciliter (g/dL), absolute neutrophil count >=1 x 10^9 cells/L, platelet count >=100x10^9 cells/L and 0% blasts in the peripheral blood. Marrow CR is defined as Bone marrow <=5% myeloblasts and decrease by >=50% over pre-treatment. Objective response rate was determined by the investigator according to international myeloma working group (IMWG) response criteria.
Time Frame: Up to 36.4 weeks
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: GSK525762 75 mg QD MDS
Number analyzed (Participants) | 16
Percentage of participants | 25 [7.3 to 52.4]

12. Primary Outcome: Part 2: Objective Response Rate Lasting at Least 4 Months (ORR4) (CTCL Cohorts)
Description: ORR4 for CTCL cohorts is defined as the percentage of participants that have achieved a CR or PR lasting at least 4 months per global response criteria and the modified severity weighted assessment tool (mSWAT). ORR4 and 95% exact confidence interval is presented.
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 1
Percentage of participants | 0 [0 to 41] | 0 [0 to 97.5]

13. Secondary Outcome: Part 1: Overall Response Rate (ORR)- Investigator Assessment
Description: ORR is defined as the percentage of participants achieving stringent complete response (sCR), very good partial response (VGPR), partial response (PR) or minimal response (MR) for multiple myeloma (MM); CR or PR for Non-Hodgkin's Lymphoma (NHL); CR, CRp, CRi or PR for Acute Myeloid Leukemia (AML); CR, MR or PR for Myelodysplastic Syndrome (MDS) using the International Working Group (IWG) response criteria and IWG response criteria in myelodysplasia.
Time Frame: Up to 86.9 weeks
Population: All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 7 | 7 | 16 | 6
Percentage of participants | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 52.2] | 0 [0 to 97.5] | 0 [0 to 60.2] | 25 [3.2 to 65.1] | 6 [0.1 to 27.3] | 0 [0 to 70.8] | 0 [0 to 36.9] | 0 [0 to 97.5] | 14 [0.4 to 57.9] | 29 [3.7 to 71.0] | 13 [1.6 to 38.3] | 17 [0.4 to 64.1]

14. Secondary Outcome: Part 1: Area Under the Concentration-time Curve (AUC) From Time Zero to 24 Hours(AUC[0-24]) and AUC Extrapolated to Infinity (AUC[0-inf]) of GSK525762 Following Single Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK525762 were collected at the indicated time points. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Week 1 Day 1: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population consisted of all participants in the All Treated Population for whom a PK sample was obtained and analyzed. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 6 | 7 | 16 | 6
Hours*nanograms per milliliter
  AUC(0-24), n=1,1,1,5,1,4,8,18,3,8,1,6,7,16, 6 | 460.48 (NA) — Geometric coefficient of variation could not be calculated for a single participant. | 1024.49 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2881.41 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2146.54 (31.68) | 3317.10 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2510.55 (71.29) | 6424.74 (22.42) | 5918.90 (52.85) | 3695.32 (62.01) | 7980.72 (45.28) | 5944.52 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 8394.69 (34.31) | 5017.96 (44.17) | 13520.57 (46.29) | 13688.54 (43.80)
  AUC(0-inf), n=1,1,1,5,1,4,7,17,3,8,1,5,7,16,5: number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 7 | 17 | 3 | 8 | 1 | 5 | 7 | 16 | 5
  AUC(0-inf), n=1,1,1,5,1,4,7,17,3,8,1,5,7,16,5 | 466.81 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1092.28 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 3054.11 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2217.32 (32.55) | 3465.49 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2546.49 (72.05) | 6951.06 (25.12) | 6214.97 (60.67) | 3874.05 (63.27) | 8248.45 (47.87) | 6032.36 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 9734.83 (29.60) | 5114.61 (44.76) | 14635.17 (52.35) | 17021.44 (35.37)

15. Secondary Outcome: Part 1: AUC(0-24) and Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) of GSK525762 Following Repeat Dose Administration
Description: Plasma samples for PK analysis of GSK525762 were collected at the indicated time points. PK parameters were calculated by standard non-compartmental analysis. AUC(0-24) represents AUC(0-tau) for repeat dose.
Time Frame: Week 2 Day 7: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 7 | 1 | 6 | 4 | 11 | 2
Hours*nanograms per milliliter
  AUC(0-24) | 476.71 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 656.93 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1855.07 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1908.18 (27.53) | 2490.25 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1702.37 (58.17) | 6271.43 (38.76) | 3576.49 (30.59) | 931.02 (53.64) | 5883.76 (48.48) | 5188.25 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 6892.57 (71.96) | 2994.24 (37.27) | 9440.98 (84.11) | 5296.46 (8.89)
  AUC(0-tau) | 476.71 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 656.93 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1855.07 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1908.18 (27.53) | 2490.25 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1702.37 (58.17) | 6271.43 (38.76) | 3576.49 (30.59) | 931.02 (53.64) | 5883.76 (48.48) | 5188.25 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 6892.57 (71.96) | 2994.24 (37.27) | 9440.98 (84.11) | 5296.46 (8.89)

16. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) and Minimum Plasma Concentration (Cmin) of GSK525762 Following Single Dose Administration
Description: Plasma samples for PK analysis of GSK525762 were collected at the indicated time points. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 6 | 7 | 16 | 6
Nanograms per milliliter (ng/mL)
  Cmax | 90.56 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 116.69 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 559.14 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 442.77 (31.83) | 513.03 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 660.79 (71.94) | 853.03 (31.1) | 1158.66 (28.58) | 813.87 (27.91) | 1728.80 (35.37) | 1248.10 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1444.42 (29.92) | 1073.51 (38.46) | 2335.99 (23.05) | 1793.39 (42.16)
  Cmin | 1.11 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 27.86 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 20.62 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 7.55 (73.07) | 21.20 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 13.25 (71.79) | 107.30 (68.40) | 50.49 (139.83) | 29.39 (47.67) | 37.92 (80.33) | 129.76 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 71.43 (112.42) | 27.89 (115.67) | 89.96 (112.80) | 138.75 (111.14)

17. Secondary Outcome: Part 1: Cmax and Cmin of GSK525762 Following Repeat Dose Administration
Description: as for outcome 16
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 7 | 1 | 6 | 4 | 11 | 2
Nanograms per milliliter (ng/mL)
  Cmax | 102.86 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 118.59 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 550.01 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 387.66 (52.41) | 557.60 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 566.59 (57.75) | 1070.32 (37.26) | 1179.42 (28.10) | 512.78 (48.37) | 1384.46 (35.35) | 1752.86 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1314.21 (58.58) | 725.29 (46.79) | 1587.25 (50.83) | 921.35 (52.16)
  Cmin | 1.47 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 5.03 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 3.92 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 7.72 (103.48) | 8.66 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2.36 (84.21) | 57.75 (82.69) | 7.03 (51.10) | 1.63 (141.42) | 14.00 (112.58) | 21.02 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 50.89 (123.69) | 4.64 (73.29) | 55.63 (163.06) | 14.96 (64.95)

18. Secondary Outcome: Part 1: Trough Concentration (Ctau) of GSK525762 Following Repeat Dose Administration
Description: as for outcome 16
Time Frame: Week 2 Day 7: Pre-dose on Days 4, 6 and 7
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 7 | 1 | 6 | 4 | 11 | 2
Nanograms per milliliter (ng/mL) | 0.91 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 3.90 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 3.76 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 4.88 (78.94) | 8.12 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 2.26 (114.63) | 32.85 (88.47) | 5.99 (41.92) | 0.03 (128.56) | 13.21 (102.35) | 2.08 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 15.77 (123.78) | 2.25 (92.05) | 42.18 (139.74) | 14.34 (68.62)

19. Secondary Outcome: Part 1: Time of Maximum Concentration (Tmax) of GSK525762 Following Single Dose Administration
Description: as for outcome 16
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 18 | 3 | 8 | 1 | 6 | 7 | 16 | 6
Hour | 0.62 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 2.00 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 1.00 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 1.00 [0.5 to 1.0] | 1.00 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 0.78 [0.4 to 2.0] | 1.56 [0.3 to 2.1] | 1.00 [0.3 to 4.1] | 1.00 [0.5 to 2.2] | 0.86 [0.5 to 2.1] | 1.28 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 1.03 [0.5 to 2.0] | 1.00 [0.3 to 1.2] | 0.92 [0.3 to 4.0] | 1.58 [0.2 to 4.1]

20. Secondary Outcome: Part 1: Tmax of GSK525762 Following Repeat Dose Administration
Description: as for outcome 16
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 7 | 1 | 6 | 4 | 11 | 2
Hour | 0.67 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 0.00 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 0.83 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 1.26 [0.5 to 2.0] | 0.50 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 0.78 [0.5 to 1.2] | 0.58 [0.5 to 2.0] | 0.50 [0.3 to 2.0] | 0.63 [0.3 to 1.0] | 0.60 [0.3 to 4.0] | 0.50 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. | 0.98 [0.5 to 2.0] | 1.06 [0.6 to 2.0] | 2.00 [0.5 to 4.0] | 2.33 [0.5 to 4.2]

21. Secondary Outcome: Part 1: Terminal Half Life (T1/2) of GSK525762 Following Single Dose Administration
Description: as for outcome 16
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 8 | 17 | 3 | 8 | 1 | 5 | 7 | 16 | 5
Hour | 4.01 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 5.75 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 6.27 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.55 [1.4 to 6.4] | 5.10 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.07 [3.5 to 4.6] | 6.48 [5.2 to 10.3] | 3.96 [2.9 to 9.3] | 5.55 [1.4 to 8.1] | 4.57 [3.3 to 6.3] | 4.15 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.75 [4.1 to 7.4] | 4.06 [3.0 to 5.8] | 5.66 [1.9 to 9.7] | 6.53 [4.7 to 7.5]

22. Secondary Outcome: Part 1: T1/2 of GSK525762 Following Repeat Dose Administration
Description: as for outcome 16
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 6 | 1 | 6 | 4 | 11 | 2
Hour | 3.68 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 5.64 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.70 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.15 [2.9 to 6.4] | 4.39 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.39 [3.2 to 5.8] | 6.48 [3.4 to 7.8] | 3.51 [3.0 to 5.3] | 1.96 [1.7 to 2.3] | 3.97 [3.1 to 5.3] | 2.54 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. | 4.98 [2.4 to 5.9] | 3.22 [2.2 to 3.7] | 5.51 [3.2 to 8.6] | 4.09 [3.8 to 4.4]

23. Secondary Outcome: Part 1: Time Invariance (RS) of GSK525762
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK525762 were collected at the indicated time points. RS was calculated by taking ratio of AUC(0-24) on Week 2 Day 7 to AUC(0-inf) on Week 1 Day 1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Week 1 Day 1: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose; Week 2 Day 7: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 5 | 1 | 4 | 3 | 10 | 2 | 7 | 1 | 7 | 4 | 11 | 1
Ratio | 1.02 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.60 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.61 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.71 (35.82) | 0.72 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.67 (18.60) | 0.98 (11.73) | 0.65 (31.37) | 0.32 (53.56) | 0.78 (46.56) | 0.86 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.91 (36.22) | 0.74 (19.36) | 0.76 (84.74) | 0.54 (NA) — Geometric coefficient of variation could not be calculated for a single participant

24. Secondary Outcome: Part 1: Accumulation Ratio (RO) of GSK525762
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK525762 were collected at the indicated time points. Accumulation ratio was calculated by taking ratio of AUC(0-24) in Week 2 Day 7 to AUC (0-24) in Week 1 Day 1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 23
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 1 | 4 | 3 | 11 | 2 | 7 | 1 | 5 | 4 | 11 | 2
Ratio | 1.04 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.64 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.64 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.74 (36.67) | 0.75 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 0.68 (17.66) | 1.06 (13.47) | 0.67 (29.24) | 0.33 (47.64) | 0.81 (45.70) | 0.87 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1.01 (33.69) | 0.75 (20.27) | 0.81 (82.45) | 0.71 (24.96)

25. Secondary Outcome: Part 2: Apparent Clearance (CL/F) of GSK525762 After Single Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK525762 were collected at the indicated time points. PK parameters were calculated by empirical Bayes estimates. GSK525762 plasma concentration-time data was analyzed by Population PK methods using a non-linear mixed-effects modelling approach.
Time Frame: Week 1 Day 1: pre-dose and at 0.5 - 2 hour, 4 - 8 hours post-dose
Population: PK Population. Given only one participant at 80 mg for single dose data, population PK analysis of combined data from 75 mg QD and 80 mg QD CTCL was more appropriate. Hence the single participant of 80 mg QD arm was included in 75 mg QD MDS arm which leads to "N" of 75 mg arm within this outcome measure is greater than overall "N" for 75 mg QD MDS & N=0 for 80 mg QC CTCL arm for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 17 | 0
Liters per hour | 11.80 (3.39) | 7.98 (3.32) |

26. Secondary Outcome: Part 2: Apparent Clearance (CL/F) of GSK525762 After Repeat Dose Administration
Description: as for outcome 25
Time Frame: Week 3 Day 1: pre-dose and at 0.5 - 2 hour, 4 - 8 hours post-dose
Population: PK Population. Given only one participant at 80 mg for single dose data, population PK analysis of combined data from 75 mg QD and 80 mg QD CTCL was more appropriate. Hence the single participant of 80 mg QD arm was included in 75 mg QD MDS arm which leads to "N=0" for 80 mg QD arm within this outcome measure.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 8 | 0
Liters per hour | 11.80 (3.39) | 9.33 (4.01) |

27. Secondary Outcome: Part 2: Apparent Central Volume of Distribution (V1/F) of GSK525762 Following Single Dose Administration
Description: as for outcome 25
Time Frame: Week 1 Day 1: pre-dose and at 0.5 - 2 hour, 4 - 8 hours post-dose
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 17 | 0
Liters | 51.5 (19.50) | 47.9 (8.01) |

28. Secondary Outcome: Part 2: Apparent Central Volume of Distribution (V1/F) of GSK525762 Following Repeat Dose Administration
Description: as for outcome 25
Time Frame: Week 3 Day 1: pre-dose and at 0.5 - 2 hour, 4 - 8 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 8 | 0
Liters | 51.5 (19.50) | 45.8 (9.92) |

29. Secondary Outcome: Part 1: AUC(0-24) and AUC[0-inf] of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: Plasma samples for PK analysis of GSK3529246 (active metabolite) were collected at the indicated time points. PK parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762.
Time Frame: Week 1 Day 1: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles). Plasma samples were not collected for analysis of GSK3529246 (active metabolite) for cohort GSK525762 5 mg QD, 10 mg QD, 20 mg QD, 40 mg QD, 60 mg QD AML, 80 mg QD, 80 mg QD AML, 120 mg QD AML.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 15 | 2 | 8 | 0 | 0 | 6 | 15 | 0
Hours*nanograms per milliliter
  AUC(0-24), n=0,0,0,5,0,1,0,15, 2,8,0,0,6,15,0 |  |  |  | 1368.11 (31.39) |  | 1891.48 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 3048.33 (22.85) | 3297.95 (68.31) | 3174.42 (40.63) |  |  | 3432.89 (39.76) | 2901.79 (52.33) |
  AUC(0-inf), n=0,0,0,5,0,1,0,10, 2,7,0,0,6,7,0: number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 10 | 2 | 7 | 0 | 0 | 6 | 7 | 0
  AUC(0-inf), n=0,0,0,5,0,1,0,10, 2,7,0,0,6,7,0 |  |  |  | 1691.75 (28.96) |  | 2013.33 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 3684.96 (28.50) | 4499.65 (72.79) | 4003.48 (42.09) |  |  | 3908.15 (41.20) | 4714.85 (48.39) |

30. Secondary Outcome: Part 1: AUC(0-24) and AUC(0-tau) of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. Pharmacokinetic parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762. AUC(0-tau) is AUC(0-24) for repeat dose.
Time Frame: Week 2 Day 7: pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed. Plasma samples were not collected for analysis of GSK3529246 (active metabolite) for cohort GSK525762 5 mg QD, 10 mg QD, 20 mg QD, 40 mg QD, 60 mg QD AML, 80 mg QD, 80 mg QD AML, 120 mg QD AML.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 2 | 7 | 0 | 0 | 4 | 10 | 0
Hours*nanograms per milliliter
  AUC(0-24) |  |  |  | 1517.96 (33.88) |  | 1922.77 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 4870.28 (46.15) | 3838.35 (37.18) | 5312.66 (45.30) |  |  | 3379.85 (44.24) | 8534.92 (43.93) |
  AUC(0-tau) |  |  |  | 1517.96 (33.88) |  | 1922.77 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 4870.28 (46.15) | 3838.35 (37.18) | 5312.66 (45.30) |  |  | 3379.85 (44.24) | 8534.92 (43.93) |

31. Secondary Outcome: Part 1: Cmax and Cmin of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. PK parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762.
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 15 | 3 | 8 | 0 | 0 | 7 | 16 | 0
Nanograms per milliliter (ng/mL)
  Cmax, n=0,0,0,5,0,1, 0,15,3,8,0,0,7,16,0 |  |  |  | 109.45 (45.38) |  | 246.12 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 239.98 (26.75) | 361.30 (54.77) | 251.73 (49.71) |  |  | 325.42 (47.17) | 201.02 (56.94) |
  Cmin, n=0,0,0,2,0,1, 0,14,3,7,0,0,6,13,0: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 14 | 3 | 7 | 0 | 0 | 6 | 13 | 0
  Cmin, n=0,0,0,2,0,1, 0,14,3,7,0,0,6,13,0 |  |  |  | 2.47 (4.29) |  | 66.39 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 18.17 (116.63) | 10.83 (161.52) | 18.45 (71.98) |  |  | 12.66 (108.08) | 14.17 (99.02) |

32. Secondary Outcome: Part 1: Cmax and Cmin of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: as for outcome 31
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 2 | 7 | 0 | 0 | 4 | 11 | 0
Nanograms per milliliter (ng/mL)
  Cmax |  |  |  | 121.83 (26.75) |  | 282.72 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 453.89 (34.07) | 500.61 (22.83) | 445.47 (52.02) |  |  | 370.67 (35.23) | 557.92 (31.81) |
  Cmin |  |  |  | 27.14 (28.38) |  | 15.18 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 66.49 (81.56) | 40.88 (45.39) | 73.60 (88.34) |  |  | 38.71 (56.34) | 116.62 (74.25) |

33. Secondary Outcome: Part 1: Trough Concentration (Ctau) of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: as for outcome 31
Time Frame: Week 2 Day 7: Pre-dose on Days 4, 6 and 7
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 2 | 7 | 0 | 0 | 4 | 10 | 0
Nanograms per milliliter (ng/mL) |  |  |  | 22.48 (36.13) |  | 13.26 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 64.57 (77.46) | 40.42 (43.96) | 76.23 (62.65) |  |  | 28.29 (94.01) | 178.76 (69.25) |

34. Secondary Outcome: Part 1: Tmax of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. Pharmacokinetic parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762.
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 30
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 15 | 3 | 8 | 0 | 0 | 7 | 16 | 0
Hour |  |  |  | 1.92 [0.9 to 4.1] |  | 0.58 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. |  | 2.10 [0.5 to 8.0] | 4.00 [2.0 to 4.2] | 3.15 [1.2 to 4.1] |  |  | 2.08 [0.3 to 4.2] | 4.03 [2.0 to 17.5] |

35. Secondary Outcome: Part 1: Tmax of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: as for outcome 34
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 30
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 2 | 7 | 0 | 0 | 4 | 11 | 0
Hour |  |  |  | 2.48 [1.0 to 4.0] |  | 0.60 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual Tmax for this single participant. |  | 1.03 [0.5 to 4.0] | 1.00 [1.0 to 1.0] | 2.05 [0.6 to 4.0] |  |  | 2.02 [1.2 to 4.1] | 4.00 [0.9 to 10.1] |

36. Secondary Outcome: Part 1: T1/2 of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: as for outcome 34
Time Frame: Week 1 Day 1: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 30
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 0 | 1 | 0 | 11 | 2 | 6 | 0 | 0 | 6 | 7 | 0
Hour |  |  |  | 9.90 [5.2 to 13.4] |  | 5.83 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant. |  | 8.66 [6.7 to 14.1] | 12.72 [11.5 to 13.9] | 8.31 [5.4 to 15.7] |  |  | 7.16 [6.3 to 9.1] | 9.23 [5.1 to 15.7] |

37. Secondary Outcome: Part 1: T1/2 of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: as for outcome 31
Time Frame: Week 2 Day 7: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 30
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 2 | 6 | 0 | 0 | 4 | 8 | 0
Hour |  |  |  | 8.24 [7.7 to 10.0] |  | 6.19 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual t1/2 for this single participant |  | 7.97 [5.7 to 12.4] | 7.39 [7.3 to 7.5] | 8.00 [5.8 to 10.5] |  |  | 6.72 [4.0 to 8.7] | 11.77 [6.9 to 23.8] |

38. Secondary Outcome: Part 1: Time Invariance (RS) of GSK3529246 (Active Metabolite)
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. RS was calculated by taking ratio of AUC(0-24) on Week 2 Day 7 to AUC(0-inf) on Week 1 Day 1. PK parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762.
Time Frame: as for outcome 23
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 8 | 1 | 6 | 0 | 0 | 4 | 6 | 0
Ratio |  |  |  | 0.92 (25.58) |  | 0.96 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 1.18 (32.33) | 0.63 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1.20 (13.74) |  |  | 1.06 (9.48) | 1.87 (57.15) |

39. Secondary Outcome: Part 1: Accumulation Ratio (RO) of GSK3529246 (Active Metabolite)
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. Accumulation ratio was calculated by taking ratio of AUC(0-24) in Week 2 Day 7 to AUC (0-24) in Week 1 Day 1. PK parameters were calculated by standard non-compartmental analysis. GSK3529246 is a metabolite of GSK525762.
Time Frame: as for outcome 23
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 9 | 1 | 7 | 0 | 0 | 4 | 9 | 0
Ratio |  |  |  | 1.18 (25.71) |  | 1.02 (NA) — Geometric coefficient of variation could not be calculated for a single participant |  | 1.61 (31.61) | 0.90 (NA) — Geometric coefficient of variation could not be calculated for a single participant | 1.56 (26.04) |  |  | 1.20 (11.50) | 3.22 (59.05) |

40. Secondary Outcome: Part 2: Apparent Clearance (CL/F) of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. GSK3529246 is a metabolite of GSK525762. PK parameters were calculated by empirical Bayes estimates. GSK3529246 plasma concentration-time data was analyzed by Population PK methods using a non-linear mixed-effects modelling approach.
Time Frame: Week 1 Day 1: pre-dose and at 0.5 - 2 hours, 4 - 8 hours post-dose
Population: PK Population. Given only one participant at 80 mg for single dose data, population PK analysis of combined data from 75 mg QD and 80 mg QD CTCL was more appropriate. Hence the single participant of 80 mg QD arm was included in 75 mg QD MDS arm which leads to "N" of 75 mg arm within this outcome measure is greater than overall "N" for 75 mg QD MDS & N=0 for 80 mg QC CTCL.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 17 | 0
Liters per hour | 16.5 (7.71) | 15.8 (6.97) |

41. Secondary Outcome: Part 2: Apparent Clearance (CL/F) of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: Plasma samples for pharmacokinetic (PK) analysis of GSK3529246 (active metabolite) were collected at the indicated time points. GSK3529246 is a metabolite of GSK525762. Pharmacokinetic parameters were calculated by empirical Bayes estimates. GSK3529246 plasma concentration-time data was analyzed by Population PK methods using a non-linear mixed-effects modelling approach.
Time Frame: Week 3 Day 1: pre-dose and at 0.5 - 2 hours, 4 - 8 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 8 | 0
Liters per hour | 15.9 (7.26) | 14.6 (8.07) |

42. Secondary Outcome: Part 2: Apparent Central Volume of Distribution (V1/F) of GSK3529246 (Active Metabolite) Following Single Dose Administration
Description: as for outcome 41
Time Frame: Week 1 Day 1: pre-dose and at 0.5 - 2 hours, 4 - 8 hours post-dose
Population: PK Population. Given only one participant at 80 mg for single dose data, population PK analysis of combined data from 75 mg QD and 80 mg QD CTCL was more appropriate. Hence the single participant of 80 mg QD arm was included in 75 mg QD MDS arm which leads to "N" of 75 mg arm within this outcome measure is greater than overall "N" for 75 mg QD MDS & N=0 for 80 mg QD CTCL.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 17 | 0
Liters | 80.0 (37.1) | 71.5 (28.4) |

43. Secondary Outcome: Part 2: Apparent Central Volume of Distribution (V1/F) of GSK3529246 (Active Metabolite) Following Repeat Dose Administration
Description: as for outcome 41
Time Frame: Week 3 Day 1: pre-dose and at 0.5 - 2 hours, 4 - 8 hours post-dose
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 8 | 0
Liters | 80.0 (37.1) | 63.4 (30.6) |

44. Secondary Outcome: Part 2: Change From Baseline in Skindex-29 Domain Scores (Emotional, Functioning and Symptoms Score) for CTCL Cohort
Description: The effects of treatment on disease-related symptoms/quality of life was assessed using the Skindex-29 Questionnaire, which inquires about how often (Never, Rarely, Sometimes, Often, All the time) during the previous 4 weeks the participant experienced the effect described in each of 29 items divided into 3 domains: Emotional (10 items), Symptoms (7 items) and Functioning (12 items). Responses to each item are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time). Skindex-29 scores were reported as three individual domain scale scores; a scale score is the mean of a participant's responses to items in a given domain. Each domain score ranges from 0 (no effect) to 100 (effect experienced all the time), higher score implies higher impact of skin disease. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline is defined is post-dose visit value minus Baseline.
Time Frame: Baseline (pre-dose Week1 Day1) and Week 3, Week 7, Week 10, Week 16 and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 6 | 1
Scores on a scale
  Emotional score, Week 3, n=6,1 | -5.83 (15.221) | 9.17 (NA) — Standard deviation could not be calculated for a single participant
  Emotional score, Week 7, n=5,0: number analyzed (Participants) | 5 | 0
  Emotional score, Week 7, n=5,0 | -19.50 (22.735) |
  Emotional score, Week 10, n=3,0: number analyzed (Participants) | 3 | 0
  Emotional score, Week 10, n=3,0 | -44.17 (26.497) |
  Emotional score, Week 16, n=3,0: number analyzed (Participants) | 3 | 0
  Emotional score, Week 16, n=3,0 | -10.00 (10.897) |
  Emotional score, Week 24, n=2,0: number analyzed (Participants) | 2 | 0
  Emotional score, Week 24, n=2,0 | -18.75 (1.768) |
  Functioning score, Week 3, n=6,1 | -1.42 (7.742) | 30.87 (NA) — Standard deviation could not be calculated for a single participant
  Functioning score, Week 7, n=5,0: number analyzed (Participants) | 5 | 0
  Functioning score, Week 7, n=5,0 | -13.37 (23.000) |
  Functioning score, Week 10, n=3,0: number analyzed (Participants) | 3 | 0
  Functioning score, Week 10, n=3,0 | -35.67 (27.820) |
  Functioning score, Week 16, n=3,0: number analyzed (Participants) | 3 | 0
  Functioning score, Week 16, n=3,0 | -13.45 (9.788) |
  Functioning score, Week 24, n=2,0: number analyzed (Participants) | 2 | 0
  Functioning score, Week 24, n=2,0 | -18.84 (11.919) |
  Symptoms score, Week 3, n=6,1 | 6.55 (24.055) | 12.50 (NA) — Standard deviation could not be calculated for a single participant
  Symptoms score, Week 7, n=5,0: number analyzed (Participants) | 5 | 0
  Symptoms score, Week 7, n=5,0 | -2.14 (18.489) |
  Symptoms score, Week 10, n=3,0: number analyzed (Participants) | 3 | 0
  Symptoms score, Week 10, n=3,0 | -29.76 (20.927) |
  Symptoms score, Week 16, n=3,0: number analyzed (Participants) | 3 | 0
  Symptoms score, Week 16, n=3,0 | -8.33 (19.670) |
  Symptoms score, Week 24, n=2,0: number analyzed (Participants) | 2 | 0
  Symptoms score, Week 24, n=2,0 | -14.29 (10.102) |

45. Secondary Outcome: Part 2: Number of Participants With Non-serious AEs and SAEs and AELDs
Description: as for outcome 1
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  Non-serious AEs | 7 | 16 | 1
  SAEs | 5 | 12 | 1
  AELD | 0 | 9 | 0

46. Secondary Outcome: Part 2: Number of Participants With Dose Reductions
Description: Number of participants with dose reductions due to any reason is presented.
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants | 6 | 7 | 0

47. Secondary Outcome: Part 2: Number of Participants With Dose Interruptions/Delays
Description: Number of participants with any dose interruptions or delays is presented.
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants | 7 | 13 | 1

48. Secondary Outcome: Part 2: Number of Participants With Grade Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: glucose, Prothrombin international normalized ratio (Pro. INR), albumin, amylase, ALT, AST, bilirubin, calcium, calcium ionized, cholesterol, creatinine, creatine kinase, lipase, potassium, magnesium, sodium, Triglycerides, ALP. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Higher grade indicates greater severity. An increase was defined as an increase relative to Baseline. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post Baseline with any grade increase is presented.
Time Frame: Up to 36.4 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  Glucose, n=7,16,1 | 6 | 14 | 1
  Pro.INR, n=4,13,0: number analyzed (Participants) | 4 | 13 | 0
  Pro.INR, n=4,13,0 | 2 | 5 |
  Albumin, n=7,16,1 | 1 | 9 | 1
  ALT, n=7,16,1 | 4 | 4 | 0
  Amylase, n=7,15,1: number analyzed (Participants) | 7 | 15 | 1
  Amylase, n=7,15,1 | 3 | 1 | 1
  AST, n=7,15,1: number analyzed (Participants) | 7 | 15 | 1
  AST, n=7,15,1 | 3 | 6 | 1
  Bilirubin, n=7,16,1 | 3 | 10 | 0
  Calcium, n=7,16,1 | 1 | 2 | 1
  Calcium Ionized, n=7,16,1 | 2 | 9 | 0
  Cholesterol, n=7,15,1: number analyzed (Participants) | 7 | 15 | 1
  Cholesterol, n=7,15,1 | 2 | 1 | 0
  Creatine Kinase, n=5,11,1: number analyzed (Participants) | 5 | 11 | 1
  Creatine Kinase, n=5,11,1 | 1 | 1 | 0
  Creatinine, n=7,16,1 | 0 | 4 | 0
  Lipase, n=7,13,1: number analyzed (Participants) | 7 | 13 | 1
  Lipase, n=7,13,1 | 2 | 2 | 1
  Potassium, n=7,16,1 | 1 | 8 | 1
  Magnesium, n=7,16,1 | 2 | 7 | 0
  Sodium, n=7,16,1 | 4 | 6 | 1
  Triglycerides, n=7,15,1: number analyzed (Participants) | 7 | 15 | 1
  Triglycerides, n=7,15,1 | 7 | 6 | 0
  ALP, n=7,16,1 | 2 | 1 | 0

49. Secondary Outcome: Part 2: Number of Participants With Grade Change From Baseline in Hematology Parameters
Description: as for outcome 6
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  Hemoglobin | 4 | 8 | 1
  Lymphocytes | 4 | 8 | 1
  Neutrophils | 2 | 7 | 0
  Platelets | 5 | 9 | 1
  Leukocytes | 1 | 6 | 0

50. Secondary Outcome: Part 2: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected to assess glucose, ketones, occult blood, urine protein. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Any increase was defined as any increase in proportional concentrations relative to Baseline. Baseline was the most recent, non-missing value prior to or on the first study treatment dose date. Data for worst-case post Baseline with any increase is presented.
Time Frame: Up to 36.4 weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 12 | 1
Participants
  Glucose, n=5,12,1: number analyzed (Participants) | 5 | 12 | 1
  Glucose, n=5,12,1 | 4 | 3 | 0
  Ketones, n=7,12,1 | 1 | 0 | 0
  Occult blood, n=7,8,1: number analyzed (Participants) | 7 | 8 | 1
  Occult blood, n=7,8,1 | 2 | 2 | 0
  Protein, n=6,11,1: number analyzed (Participants) | 6 | 11 | 1
  Protein, n=6,11,1 | 0 | 7 | 0

51. Secondary Outcome: Part 2: Number of Participants With Worst Case Vital Signs Results Relative to Baseline: Pulse Rate and Body Temperature
Description: as for outcome 8
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  Pulse rate, To Low | 2 | 0 | 0
  Pulse rate, To Normal or No change | 3 | 9 | 0
  Pulse Rate, To High | 3 | 7 | 1
  Temperature, To Low | 1 | 0 | 0
  Temperature, To Normal or No Change | 5 | 13 | 1
  Temperature, To High | 1 | 3 | 0

52. Secondary Outcome: Part 2: Number of Participants With Increase to Grade 3 From Baseline in Vital Signs: DBP and SBP
Description: as for outcome 9
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  DBP | 0 | 0 | 0
  SBP | 3 | 1 | 1

53. Secondary Outcome: Part 2: Number of Participants With Worst-case Post-Baseline Abnormal Electrocardiogram (ECG) Findings (Investigator Reading)
Description: as for outcome 10
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Participants
  Abnormal-Clinically significant | 0 | 1 | 0
  Abnormal-Not Clinically significant | 6 | 11 | 1

54. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: PFS defined as interval of time(in months) between date of first dose & earlier of date of disease progression & date of death due to any cause.Progression is participants(pt's)with MDS & with <5% blasts:>=50% increase in blasts to>5% blasts/pt's with 5-10% blasts:>=50% increase to >10% blasts, for pt's with 10-20% blasts:>=50% increase to >20% blasts,for pt's with 20%-30% blasts:>=50% increase to >30% blasts, for CTCL progression is >=25% increase in skin disease from Baseline/new tumors (T3[1 or more tumors(>=1cm diameter]) in pt's with T1(Limited patches,papules&/or plaques covering <10% of the skin surface;may further stratify into T1a [patch only] versus T1b [plaque+-patch]),T2(Patches,papules/plaques covering >=10% of skin surface;may further stratify into T2a[patch only]versus T2b [plaque+-patch]) orT4(Confluence of erythema covering >=80% body surface area) only skin disease/loss of response in those with CR/PR, increase of skin score of > sum of nadir +50% Baseline score.
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Months | 8.15 [3.48 to NA] — Third quartile could not be calculated | 2.00 [1.45 to 3.48] | NA [NA to NA] — No event occurred for single participant hence Median and Inter-quartile range could not be calculated

55. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: Duration of response is defined as the time from the first documented evidence response (CR or PR lasting 4 months for CTCL; and CR, marrow CR, CRp, Cri or PR for MDS) until the first documented disease progression or death due to any cause. Median and inter-quartile range (first quartile and third quartile) of duration of response are presented.
Time Frame: Up to 36.4 weeks
Population: All treated Population. Only those participants with data available at the specified data points were analyzed. Participants with incomplete response rates were excluded from the analysis hence N=0 for 60 mg QD and 80 mg QD CTCL arms.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 0 | 4 | 0
Months |  | 3.29 [3.29 to 3.29] |

56. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS is defined as the interval of time (in months) between the date of first dose and the date of death due to any cause. Median and inter-quartile range (first quartile and third quartile) of overall survival are presented.
Time Frame: Up to 36.4 weeks
Population: All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 7 | 16 | 1
Months | NA [NA to NA] — Median and inter-quartile range was not reached. | 5.85 [1.46 to 16.10] | NA [NA to NA] — No event occurred for single participant hence Median and Inter-quartile range could not be calculated.

57. Other Pre Specified Outcome: Part 2: Time to Progression (TTP) for Participants With MM
Description: Time to Progression was planned to be analyzed.
Time Frame: Up to 36.4 weeks
Population: All Treated Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 0 | 0 | 0

58. Other Pre Specified Outcome: Part 1: Changes in Cardiac QT Duration Corrected for Heart Rate by Fridericia's Formula (QTcF) and Other Safety Parameters in Relation to GSK525762 PK Concentrations
Description: Changes in QTcF and other safety parameters in relation to GSK525762 PK concentrations was planned to be analyzed.
Time Frame: Up to 86.9 weeks
Population: All Treated Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

59. Other Pre Specified Outcome: Part 1: Number of Participants With Dose /Exposure Markers Related Change in Molecular Markers in Tumor Tissue and/or Peripheral Blood Samples
Description: Number of participants with dose /exposure markers related change in molecular markers (e.g. gene transcription and/or expression of proteins regulated by Bromodomain [BRD] proteins) in tumor tissue and/or peripheral blood samples were planned to be analyzed.
Time Frame: Up to 86.9 weeks
Population: All Treated Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

60. Other Pre Specified Outcome: Part 2: Plasma Concentrations of GSK525762 in Relationship With Safety and Efficacy Parameters Derived From Pharmacokinetic/Pharmacodynamic (PK/PD) Model
Description: Plasma concentrations of GSK525762 in relationship with safety and efficacy parameters derived from PK/PD model was planned to be analyzed.
Time Frame: Up to 36.4 weeks
Population: PK Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 0 | 0 | 0

61. Other Pre Specified Outcome: Part 2: Number of Participants With Dose /Exposure Markers Related Change in Molecular Markers in Tumor Tissue and/or Peripheral Blood Samples
Description: Number of participants with dose /exposure markers related change in molecular markers (e.g. gene transcription and/or expression of proteins regulated by Bromodomain proteins) in tumor tissue and/or peripheral blood samples were planned to be analyzed.
Time Frame: Up to 36.4 weeks
Population: All Treated Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 2: GSK525762 60 mg QD CTCL | Part 2: GSK525762 75 mg QD MDS | Part 2: GSK525762 80 mg QD CTCL
Number analyzed (Participants) | 0 | 0 | 0

62. Other Pre Specified Outcome: Part 1: Overall Survival (OS)
Description: Overall survival (defined as the interval of time in months between the date of first dose and the date of death due to any cause) was planned to be analyzed.
Time Frame: Up to 86.9 weeks
Population: All Treated Population. This was an other pre-specified outcome measure. Data was not analyzed and reported.
Arm/Group | Part 1: GSK525762 5 mg QD | Part 1: GSK525762 10 mg QD | Part 1: GSK525762 20 mg QD | Part 1: GSK525762 30 mg QD MM | Part 1: GSK525762 40 mg QD | Part 1: GSK525762 40 mg QD MM | Part 1: GSK525762 60 mg QD AML | Part 1: GSK525762 60 mg QD NHL | Part 1: GSK525762 60 mg QD MM | Part 1: GSK525762 75 mg QD AML | Part 1: GSK525762 80 mg QD | Part 1: GSK525762 80 mg QD AML | Part 1: GSK525762 80 mg QD NHL | Part 1: GSK525762 100 mg QD AML | Part 1: GSK525762 120 mg QD AML
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious and serious adverse events were collected from the start of study treatment until 28 days following discontinuation of study treatment (up to 86.9 weeks for Part 1 and up to 36.4 weeks for Part 2)
Description: All-cause mortality, non-serious AEs and SAEs were collected in All Treated population.
Groups:
- GSK525762 5 MG QD: Participants were administered once daily oral dose of 5 milligrams (mg) GSK525762.
- GSK525762 10 MG QD: Participants were administered once daily oral dose of 10 mg GSK525762.
- GSK525762 20 MG QD: Participants were administered once daily oral dose of 20 mg GSK525762.
- GSK525762 30 MG QD MM: Participants with multiple myeloma (MM) were administered once daily oral dose of 30 mg GSK525762.
- GSK525762 40 MG QD: Participants were administered once daily oral dose of 40 mg GSK525762.
- GSK525762 40 MG QD MM: Participants with MM were administered once daily oral dose of 40 mg GSK525762.
- GSK525762 60 MG QD AML: Participants with Acute Myeloid Leukemia (AML) were administered once daily oral dose of 40 mg GSK525762.
- GSK525762 60 MG QD NHL: Participants with Non-Hodgkin's Lymphoma (NHL) were administered once daily oral dose of 60 mg GSK525762.
- GSK525762 60 MG QD MM: Participants with MM were administered once daily oral dose of 60 mg GSK525762.
- GSK525762 75 MG QD AML: Participants with AML were administered once daily oral dose of 75 mg GSK525762.
- GSK525762 80 MG QD: Participants were administered once daily oral dose of 80 mg GSK525762.
- GSK525762 80 MG QD AML: Participants with AML were administered once daily oral dose of 80 mg GSK525762.
- GSK525762 80 MG QD NHL: Participants with NHL were administered once daily oral dose of 80 mg GSK525762.
- GSK525762 100 MG QD AML: Participants with AML were administered once daily oral dose of 100 mg GSK525762.
- GSK525762 120 MG QD AML: Participants with AML were administered once daily oral dose of 120 mg GSK525762.
- GSK525762 60 MG QD CTCL: Participants Cutaneous T cell lymphoma (CTCL) were administered once daily oral dose of 60 mg GSK525762.
- GSK525762 75 MG QD MDS: Participants with Myelodysplastic Syndrome (MDS) were administered once daily oral dose of 75 mg GSK525762.
- GSK525762 80 MG QD CTCL: Participants CTCL were administered once daily oral dose of 80 mg GSK525762.
Arm/Group | GSK525762 5 MG QD | GSK525762 10 MG QD | GSK525762 20 MG QD | GSK525762 30 MG QD MM | GSK525762 40 MG QD | GSK525762 40 MG QD MM | GSK525762 60 MG QD AML | GSK525762 60 MG QD NHL | GSK525762 60 MG QD MM | GSK525762 75 MG QD AML | GSK525762 80 MG QD | GSK525762 80 MG QD AML | GSK525762 80 MG QD NHL | GSK525762 100 MG QD AML | GSK525762 120 MG QD AML | GSK525762 60 MG QD CTCL | GSK525762 75 MG QD MDS | GSK525762 80 MG QD CTCL
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 4/5 | 0/1 | 3/4 | 7/8 | 12/18 | 2/3 | 8/8 | 1/1 | 7/7 | 6/7 | 15/16 | 6/6 | 1/7 | 13/16 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 4/5 | 0/1 | 3/4 | 6/8 | 12/18 | 2/3 | 8/8 | 1/1 | 6/7 | 7/7 | 14/16 | 6/6 | 5/7 | 12/16 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 5/5 | 1/1 | 4/4 | 8/8 | 18/18 | 3/3 | 8/8 | 1/1 | 7/7 | 7/7 | 16/16 | 6/6 | 7/7 | 16/16 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK525762 5 MG QD (N=1) | GSK525762 10 MG QD (N=1) | GSK525762 20 MG QD (N=1) | GSK525762 30 MG QD MM (N=5) | GSK525762 40 MG QD (N=1) | GSK525762 40 MG QD MM (N=4) | GSK525762 60 MG QD AML (N=8) | GSK525762 60 MG QD NHL (N=18) | GSK525762 60 MG QD MM (N=3) | GSK525762 75 MG QD AML (N=8) | GSK525762 80 MG QD (N=1) | GSK525762 80 MG QD AML (N=7) | GSK525762 80 MG QD NHL (N=7) | GSK525762 100 MG QD AML (N=16) | GSK525762 120 MG QD AML (N=6) | GSK525762 60 MG QD CTCL (N=7) | GSK525762 75 MG QD MDS (N=16) | GSK525762 80 MG QD CTCL (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (9) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 2 (2) | 5 (11) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucormycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | GSK525762 5 MG QD (N=1) | GSK525762 10 MG QD (N=1) | GSK525762 20 MG QD (N=1) | GSK525762 30 MG QD MM (N=5) | GSK525762 40 MG QD (N=1) | GSK525762 40 MG QD MM (N=4) | GSK525762 60 MG QD AML (N=8) | GSK525762 60 MG QD NHL (N=18) | GSK525762 60 MG QD MM (N=3) | GSK525762 75 MG QD AML (N=8) | GSK525762 80 MG QD (N=1) | GSK525762 80 MG QD AML (N=7) | GSK525762 80 MG QD NHL (N=7) | GSK525762 100 MG QD AML (N=16) | GSK525762 120 MG QD AML (N=6) | GSK525762 60 MG QD CTCL (N=7) | GSK525762 75 MG QD MDS (N=16) | GSK525762 80 MG QD CTCL (N=1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 3 (6) | 7 (8) | 0 (0) | 4 (4) | 1 (2) | 4 (6) | 3 (3) | 11 (15) | 3 (3) | 2 (2) | 11 (14) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 6 (7) | 2 (2) | 4 (4) | 0 (0) | 6 (6) | 2 (2) | 8 (10) | 3 (4) | 2 (2) | 11 (12) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 11 (11) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 6 (6) | 1 (1) | 3 (4) | 6 (6) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (8) | 7 (7) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 7 (8) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 8 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 2 (2) | 0/0 (0) | 0 (0) | 1 (1) | 0 (0) | 1/1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 3 (3) | 1/1 (1) | 0/0 (0) | 0/0 (0) | 0/0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT01943851/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT01943851/SAP_001.pdf